CLINICAL TRIAL: NCT05266755
Title: Hospital Readmission After HIPr Fracture. Impact of a Territorial Fracture Liason Service
Acronym: FLSSantPau
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-FLS-2021-114
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Multicenter clinical trial. Adult patients who consult the Hospital Emergency Department (ED) of the Hospital de la Santa Creu i Sant Pau (HSCSP) for an FxF PSM as a primary or secondary diagnosis will be selected and will be randomized with a 1:1 distribution to be included in the FLS -CTSPau (intervention group) or to receive usual care (control group). The result of the intervention will be evaluated in terms of health outcomes (re-consultations, hospital readmissions and quality of life).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patiens who will receive stanrdar care after hip fracture (Placebo Comparator): All the patients who will be on surgery after a hip fracture will receive after the hospital discharge the standar following we are doing now in our hospital
  Interventions: Other: Fracture Territorial Liaison Service afert a Hip fracture
- Patiens who will receive FLS following after the hip fracture (Active Comparator): All the patients who will be on surgery after a hip fracture will receive after the hospital discharge a FLS following, multidisciplinary, with a web and mobile app aplication
  Interventions: Other: Fracture Territorial Liaison Service afert a Hip fracture

INTERVENTIONS:
Other: Fracture Territorial Liaison Service afert a Hip fracture — Give a diferent than the current one way of follow up to the patients with hip fracture

SUMMARY:
The International Osteoporosis Foundation (IOF) and the American Society for Bone Research and Mineral Metabolism recommend the creation and implementation of fracture coordination services (FLS) as the most efficient way to address the problem. FLS has emerged as a new clinical approach that uses coordinated, multidisciplinary care to improve post-fracture outcomes and reduce recurrent fractures. It is a multidisciplinary and protocolized care model that must guarantee:

1. Identify fragility fractures and people at risk for a fracture
2. Fracture risk assessment
3. Indication for treatment or referral
4. Improvement in therapeutic compliance
5. Reduce the risk of falls It is known that patients who have undergone a FLS model (vs no FLS), have lower mortality, lower risk of fracture, with a reduction of 35% and 56%, respectively, during two years of follow-up. One of the most important objectives of the FLS is the proper recognition and treatment of osteoporosis (OP) in patients with fragility fractures. A major problem is the lack of adherence to treatment for OP, and inclusion in an FLS program increases the prescription of bisphosphonates from 17.9% to 76%. In addition, a specific follow-up program means that 73% of patients followed by FLS continue to undergo anti-resorptive treatment after 2 years of having suffered a femur fracture.

DETAILED DESCRIPTION:
Hypothesis After a femur fracture due to fragility, upon discharge from surgery at the Hospital de la Santa Creu i Sant Pau, including patients in a regional FLS program will make it possible to complete the study of the patient with fracture, improve adherence to treatment of OP (secondary prevention), and obtain better functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* All hip fractures older than 65 years

Exclusion Criteria:

* Politraumatic fractures
* Metastasic fractures

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Deaths | 1 year after discharge
  % of Number of deaths after 1st year o follow up
Number of Falls | 1 year after discharge
  Number of Falls 1st year o follow up
Percentage of patients with adequated Osteoporotic treatment | 1 year after discharge
  Percentage of patients with adequated osteoporotic treatment

SECONDARY OUTCOMES:
Barthel at the end of follow up | 1 year after discharge
  Compare Barthel after hospital discharge with the end of follow up barthel. Minimum is 0 maximum is 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordi Martin Marcuello, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided